CLINICAL TRIAL: NCT04181658
Title: The Feasibility and Effectiveness of Combining Non-invasive Brain Stimulation and Physical Therapy to Improve Gait and Balance in Older Adults at Risk of Falling
Brief Title: The Brain Stimulation and Physical Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2019-24
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Fall; Gait, Unsteady; Aging; Accidental Fall
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS and Physical Therapy (Experimental): This arm combines tDCS and Physical Therapy intervention. The real tDCS will be delivered before each physical therapy visit for up to 10 combined sessions. The tDCS montage was designed to target the left dorsal lateral prefrontal cortex (DLPFC) for around 20 minutes. The direct current delivered by any electrode will not exceed 2.0 milliamp(mA) and the total amount of current from all electrodes will not exceed 4 mA.
  Interventions: Other: Real tDCS and Physical Therapy
- Sham stimulation and Physical Therapy (Sham Comparator): This arm combines sham stimulation and Physical Therapy intervention. The sham stimulation will be delivered before each physical therapy visit for up to 10 combined sessions. We will use an active sham stimulation in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session. This montage was designed to deliver currents not significantly influence their cortical tissue, but still, mimic the cutaneous sensations induced by tDCS over the same brain site (i.e. left DLPFC).
  Interventions: Other: Sham stimulation and Physical Therapy

INTERVENTIONS:
Other: Real tDCS and Physical Therapy — The participant will receive 20-minute sessions of real tDCS before each physical therapy visit for up to 10 combined sessions, over approximately 6 weeks.
  Other Names: Real tDCS + PT
  Arms: Real tDCS and Physical Therapy
Other: Sham stimulation and Physical Therapy — The participant will receive 20-minute sessions of sham stimulation before each physical therapy visit for up to 10 combined sessions, over approximately 6 weeks.
  Other Names: Sham stimulation + PT
  Arms: Sham stimulation and Physical Therapy

SUMMARY:
This pilot work will determine the feasibility of tDCS intervention as an effective adjunct intervention to PT aimed at improving gait, balance, and mobility in older adults at risk of falling.

DETAILED DESCRIPTION:
Falls are correlated with both physical and cognitive declines in older adults. Recurrent fallers and those at high risk of falls are often referred to physical therapy (PT) for gait and balance training. Although physical therapists are aware of the importance of cortical control of gait and balance, there is no available tool to directly yet non-invasively intervene brain in the clinical setting.

Transcranial direct current stimulation (tDCS) is a noninvasive and safe mean of modulating the excitability of specific brain regions and their connected neural networks. Our group and others have shown that tDCS intervention designed to facilitate the excitability of the left dorsal lateral prefrontal cortex (DLPFC) improves numerous aspects of executive function related to mobility in older adults. However, no studies to date have assessed the feasibility and effectiveness of applying tDCS as an adjunct to PT to improve gait and balance within the geriatric rehabilitation setting.

This study aims to 1) assess the feasibility of implementing tDCS prior to each of their first 10 PT sessions, and 2) gather estimates of variability in outcomes related to gait, balance, cognition, and quality of life over time within older adults referred to PT for recurrent falls.

ELIGIBILITY:
Inclusion Criteria:

* Ages 65 years old and above
* Admitted to Physical Therapy for gait and balance training due to the high risk of falls

Exclusion Criteria:

* Inability to stand or walk unassisted for 60 seconds
* Severe cognitive impairment defined as a Montreal Cognitive Assessment (MoCA) score < 18
* Any unstable medical condition
* Any unstable psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* Active cancer for which chemo/radiation therapy id being received
* Significant vision and hearing problems that cannot be corrected with visual and hearing aids
* Contraindications to tDCS, including seizure within the past two years, use of neuro-active drugs, the risk of metal objects in the brain, implanted medical devices, or the presence of dermatological conditions such as eczema on the scalp.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Screening to enrollment ratio (%, 0-100, higher ratio means a better outcome) | The whole data collection period (~ 6 months for the whole study)
  The number of screenings needed to enroll one participant
Intervention adherence rate (%, 0-100, higher ratio means a better outcome) | The whole data collection period (~ 6 months for the whole study)
  Number of tDCS sessions completed
Adherence rate (%, 0-100, higher ratio means a better outcome) | The whole data collection period (~ 6 months for the whole study)
  The portion of enrolled participants who complete and adhere to the intervention who complete and adhere to the intervention
Side effects | The whole data collection period (~ 6 months for the whole study)
  The number, type, severity and duration of reported side effects
Change from baseline in the dual task cost to gait speed (reduced dual task cost after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in the degree to which performing a secondary cognitive task diminishes gait speed
Change from baseline in the dual task cost to standing postural sway speed (reduced dual task cost after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in the degree to which performing a secondary cognitive task diminishes the control of standing posture.
Change from baseline in Trail Making Test B - A (reduced time after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in cognitive executive function

SECONDARY OUTCOMES:
Change from baseline in gait speed (increased value after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in gait speed
Change from baseline in gait variability (reduced value after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in gait speed
Change from baseline in gradual-onset continuous performance test (gradCPT) ( increased accuracy after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in cognitive sustained attention
Change from baseline in Timed Up-and-Go (TUG) (reduced time after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in overall mobility function
Change from baseline in Montreal Cognitive Assessment (MoCA) total score (increased score after intervention means a better outcome) | Before and after the intervention (~ 6 weeks per participant)
  The change from baseline in global cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: On-Yee Lo, PhD, Principal Investigator — Hebrew Rehabilitation Center
Locations (1):
- Hebrew Rehabilitation Center, Boston, Massachusetts, United States